CLINICAL TRIAL: NCT00320294
Title: A Randomized Trial of Irinotecan, Leucovorin, 5-FU (ILF) Versus ILF Plus Cisplatin (PILF) Combination Chemotherapy in Patients With Advanced Gastric Cancer
Brief Title: ILF With/Without Cisplatin for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMO-GI-52
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2007-03-12 (Estimated); Status verified 2007-03

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan; Cisplatin

INTERVENTIONS:
Drug: irinotecan
Drug: cisplatin

SUMMARY:
To compare the combination of irinotecan, leucovorin and 5-FU (ILF) with ILF plus cisplatin (PILF) as first-line chemotherapy in patients with measurable metastatic gastric cancer.

DETAILED DESCRIPTION:
Irinotecan, in combination with 5-FU or cisplatin, clearly demonstrated efficacy against gastric cancer. A previous randomized study of ILF regimen versus IP in patients with AGC showed that the ILF produced an overall response rate of 42% and a median survival of 10.7 months, which were significantly better than the results with IP regimen [Pozzo C, et al. Ann Oncol 2004]. However, since cisplatin is still considered one of the key drugs for the treatment of gastric cancer, a combination of these four drugs (irinotecan, leucovorin, FU and cisplatin) seemed to be a promising strategy for advanced AGC. We desinged this randomized phase II study to compare the combination of irinotecan, leucovorin and 5-FU (ILF) with ILF plus cisplatin (PILF) as first-line chemotherapy in patients with measurable metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric adenocarcinoma
* Advanced, metastatic or recurrent
* ECOG performance status 0 to 2
* No prior chemotherapy
* Measurable or evaluable indicator lesion(s)
* Normal marrow, hepatic and renal functions
* Provision of written informed consent

Exclusion Criteria:

* Active infection, bleeding or severe comorbidities
* Pregnant or breastfed women
* Active CNS metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2005-02; Study Completion 2007-03

PRIMARY OUTCOMES:
Objective response rate
Safety

SECONDARY OUTCOMES:
Progression-free survival
Overall survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Park SH, Nam E, Park J, Cho EK, Shin DB, Lee JH, Lee WK, Chung M, Lee SI. Randomized phase II study of irinotecan, leucovorin and 5-fluorouracil (ILF) versus cisplatin plus ILF (PILF) combination chemotherapy for advanced gastric cancer. Ann Oncol. 2008 Apr;19(4):729-33. doi: 10.1093/annonc/mdm502. Epub 2007 Dec 13. PMID 18083691